CLINICAL TRIAL: NCT00841737
Title: Evaluation of the Effectiveness and Efficiency of a Psychoeducational Group Sessions Intervention Program in the Depressive Episode Realized by Primary Health Care Center Nurses in Barcelona City.
Brief Title: Evaluation of a Psychoeducation Group Program for Mild/Moderate Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Hospital Universitari Vall d'Hebron Research Institute (Other); Centre d'Higiene Mental Les Corts (Other)
Responsible Party: Rocio Casañas, Barcelona Primary Care Area . Catalan Health Institute (Institut Catala de la Salut (ICS)).
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI07/90712
Record Dates: First submitted 2009-02-03; First posted 2009-02-11 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Depressive Disorders
Keywords: Depressive Disorders;; Primary Health Care;; Nurses;; Health education.
MeSH Terms: conditions — Depressive Disorder; Health Education | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychoeducational group intervention (Experimental): Psychoeducational group received weekly a psychoeducational intervention during a period of 12 weeks run by a nurses.
  Interventions: Other: Psychoeducational group
- Control group (Active Comparator): Individual conventional care
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Psychoeducational group — The intervention group receive weekly a psychoeducational group during 12 weeks run by 2 nurses. The program have a structures contend.
  Other Names: Psychoeducational group;; Depression group intervention.
  Arms: Psychoeducational group intervention
Other: Control Group — In the control group the depression is treated as usual with the conventional treatment.
  Other Names: conventional treatment group;; usual care group
  Arms: Control group

SUMMARY:
The purpose of this study is to compare the effectiveness and efficiency of doing a psychoeducational group program and the conventional treatment versus individual conventional care in patients with a mild/moderate depression disorder,in urban primary healthcare centers in Barcelona city.

DETAILED DESCRIPTION:
Nowadays, the depression is one of the public health major issues, this is because of its prevalence and its economic and social repercussions. It is fundamental for the Primary Care to assume the management of these health problems.

Design:A randomised controlled trial of two groups (intervention and control), longitudinal and prospective.

Population of study: The subjects of the study are patients of 20 to 65 years old attended in 8 urban primary healthcare centers of Barcelona city, identified by the general practitioners and nurses with diagnosis of mild/moderate depression disorder according to the BDI scale.

The intervention group receive weekly a psychoeducational group program during 12 weeks run by 2 nurses. The program have a structured content where patient is educated about the illness, pharmacological treatment, the adherence to treatment, diet and physical exercise, problem solving, and cognitive-behavioral therapy.

In the control group the depression in treated as usual with the conventional care.

Measure's tool: The evolution of patients will be monitoring up to 1 year after the inclusion by a individual interview (the first visit and 3,6 and 9 months).The Beck Depression inventory (BDI) is a self-administered questionnaire that measure the symptomatology and severity of the depression.

The analysis variables are: patient's quality of life (EuroQoL-5D scale) ,clinical variables of the patient, pharmacological prescription, anxiolytics and antidepressants consumption , sociodemographic, number of visits to primary healthcare center, number of days of labour lost and cost.

ELIGIBILITY:
Inclusion Criteria:

* Beck Depression Inventory(BDI)>10 and <30.
* Diagnosis of mild/moderate depressive disorders.
* Signed the Informed Consent.

Exclusion Criteria:

* Patients diagnosed of severe mental psychiatric disorder,
* Patients diagnosed of a major depressive disorders,
* Patients with acute illness or near-terminal medical illness,
* using secondary mental health services,
* suicidal ideation or intentions,
* don't speak and understand spanish or/and catalan language,
* sensory or cognitive disabilities,
* illiteracy,
* does not know or not give consent to participate in the study,
* temporary residents.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
To measure the symptomatology of the depression by Beck Depression Inventory (BDI) It's a self-administered questionnaire with 21 items (multiple-choice)to measure the intensity, severity and depth of depression. | First visit and 3, 6 and 9 months.

SECONDARY OUTCOMES:
To measure the patient's quality of life by the EuroQoL questionnaire; number of visits to primary health care center( doctor and nurse); number of days of labour lost; pharmacological prescription; antidepressant and anxiolytics consumption. | First visit and 3,6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Casañas, Psychologist, Principal Investigator — Barcelona Primary Care Area. Catalan Health Institute (ICS)
Locations (2):
- Spain (2):
  - Primary Health Care . Catalan Health Institute (ICS), Barcelona, Barcelona
  - Primary health care. Catalan Health Institute (ICS), Barcelona, Barcelona

REFERENCES:
- [Derived] Casanas R, Catalan R, del Val JL, Real J, Valero S, Casas M. Effectiveness of a psycho-educational group program for major depression in primary care: a randomized controlled trial. BMC Psychiatry. 2012 Dec 18;12:230. doi: 10.1186/1471-244X-12-230. PMID 23249399